CLINICAL TRIAL: NCT05976386
Title: A Randomized, Open-label, Parallel Design, Single Dose Study to Compare the Pharmacokinetics of New and Current Dupilumab Drug Products Subcutaneously Administered in Healthy Adults
Brief Title: Single Dose Comparability Study of New and Current Dupilumab Drug Products Subcutaneously Administered in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKM17324; U1111-1266-7002 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- New dupilumab product (Experimental): A single subcutaneous injection on Day 1
  Interventions: Drug: Dupilumab (SAR231893)
- Current dupilumab product (Active Comparator): A single subcutaneous injection on Day 1
  Interventions: Drug: Dupilumab (SAR231893)

INTERVENTIONS:
Drug: Dupilumab (SAR231893) — Injection solution Subcutaneous
  Other Names: REGN668

SUMMARY:
This is a parallel group, treatment, Phase 1, open-label, 2-arm study to demonstrate pharmacokinetic comparability between subcutaneous (SC) single dose of new dupilumab product and SC single dose of current dupilumab product in male and female healthy participants aged 18 to 65 years.

The estimated duration is up to 21 days of screening period, followed by the treatment day with a follow-up treatment period of 42 days until the end of study (EOS) visit. Total duration from screening to EOS will be 64 days maximum.

DETAILED DESCRIPTION:
Duration per participant is up to 64 days

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, between 18 and 65 years of age, inclusive.
* Body weight between 65.0 and 95.0 kg, inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Having given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

* Presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month).
* Blood donation, any volume, within 2 months before inclusion.
* Presence or history of drug or biologic hypersensitivity, or allergic disease diagnosed and treated by a physician (excluding seasonal allergy).
* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day on a regular basis).
* Smoking regularly and unable to stop smoking during the inpatient portion of the study (occasional smoker can be enrolled).
* If female, pregnancy (defined as positive β-human chorionic gonadotropin (HCG) blood test) or breastfeeding.
* Any biologics (antibody or its derivatives) given within 4 months before inclusion or within 5 half-lives (whichever takes longer).
* Participation in any previous clinical trial of dupilumab.
* Participation in any clinical research study evaluating another investigational drug or therapy in which the inclusion visit for the current study will be within 30 days of receiving the drug or 5 elimination half-lives (whichever is longer).
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Maximum serum concentration of functional dupilumab (Cmax) | Pre-dose on Day 1 up to Day 43
Area under the serum concentration versus time curve from time zero to the real time of last measurable concentration (AUClast) | Pre-dose on Day 1 up to Day 43

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Day 1 up to Day 43

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami-Site Number:8400001, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PKM17324 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25328&tenant=MT_SNY_9011